CLINICAL TRIAL: NCT05439187
Title: Risk Factors of Venous Thromboembolism After Incisional Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Igor Zolotukhin, Professor, Pirogov Russian National Research Medical University
Other Study IDs: 140-14/22
Record Dates: First submitted 2022-05-23; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Incisional Hernia; Venous Thromboembolism
Keywords: hernia repair; thromboprophylaxis
MeSH Terms: conditions — Incisional Hernia; Venous Thromboembolism | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hernia repair — Open or laparoscopic hernia repair with mesh placement.
  Other Names: thromboprophylaxis

SUMMARY:
Aim of our study is to find frequency and risk factors for venous thromboembolism development in patients who underwent surgery for incisional ventral hernia. There were 240 patients enrolled in our retrospective observational cohort study. Included patients were operated for incisional hernia in Saveljev University Surgery Clinic from January 2018 to December 2019. Compression duplex ultrasound of lower legs veins was performed in 2-4 days after surgery for all participants. The primary endpoint was the occurrence of the venous thromboembolism event, including pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* operated for incisional hernia in Saveljev University Surgery Clinic No Exclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of Saveljev University Surgery Clinic, Moscow
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
venous thromboembolism | was performed with median 3 days (min 1 day, max 7 days, interquartile range 2-4 days) after surgery
  Screening ultrasound in the postoperative period was aimed at looking for signs of deep vein thrombosis. The imaged vessels included the common femoral, great saphenous, superficial femoral, deep femoral, popliteal, posterior tibial, and peroneal veins of both lower extremities. The presence of a thrombotic process in the vein was evidenced by the rigidity of its walls during compression by the sensor, the presence of hyperechoic inclusions, and the impossibility of visualizing blood flow during color mapping.

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Russia